CLINICAL TRIAL: NCT03497260
Title: Fructose to Reduce Exercise-associated Hypoglycaemia in Individuals With Type 1 Diabetes Treated With Insulin Degludec: Questioning a Paradigm and Offering a Novel Strategy
Brief Title: Fructose in Exercising Individuals With Type 1 Diabetes Using Insulin Degludec
Acronym: FruDeg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: FruDeg
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Type 1 Diabetes Mellitus; Diabetes Complications
Keywords: Type 1 Diabetes, Fructose, Exercise, Hypoglycaemia, Degludec
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Complications; Motor Activity; Hypoglycemia | interventions — Fructose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fructose in water first, water only second (Experimental): Intake of 20 g of fructose dissolved in 200 ml of tap water at first visit; intake of 200 ml of tap water at second visit
  Interventions: Dietary Supplement: Fructose; Other: Plain water
- Water only first, Fructose in water second (Experimental): Intake of 200 ml of tap water at first visit; intake of 200 ml of 20 g of fructose dissolved in 200 ml of tap water at second visit
  Interventions: Dietary Supplement: Fructose; Other: Plain water

INTERVENTIONS:
Dietary Supplement: Fructose — Intake of 20 g of fructose dissolved in 200 ml of tap water within 5 minutes 30 minutes prior to exercise.
Other: Plain water — Intake of 200 ml of tap water within 5 minutes 30 minutes prior to exercise.

SUMMARY:
To determine and compare the time-to-hypoglycaemia (defined as plasma glucose <3.9mmol/L) in individuals with type 1 diabetes treated with ultra-Long acting insulin degludec during aerobic exercise with or without prior ingestion of a single oral fructose load.

DETAILED DESCRIPTION:
Glycaemic control remains complex and demanding during exercise for type 1 diabetes (T1D) patients. Traditional treatment guidelines for exercise emphasizing the reduction of insulin doses and/or ingestion of additional carbohydrates are of limited applicability for patients treated with ultra-long acting basal insulin analogues. Dose reductions may require two to three days for modern basal insulin analogues in order to achieve an adapted steady state, hereby increasing the risk of inadequate insulin-following exercise. If T1D patients engage in recreational exercise - as recommended by every international treatment guideline - current treatment strategies may simply not be sufficient.

As a consequence for patients treated with modern basal insulin analogues, it seems more adequate not to modify insulin doses but to apply alternative strategies for recreational exercise. The ingestion of fructose, an insulin-independent carbohydrate, which increases lipid oxidation but attenuates the dependency on carbohydrates may offer a novel strategy. Up to date, only preliminary data for fructose have been produced regarding clinical effectiveness and underlying mechanisms in the prevention of hypoglycaemia. The present comprehensive study aims to investigate the clinical efficacy, feasibility, and safety of a pre-exercise oral fructose load without modification of insulin degludec in T1D patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes as defined by the World Health Organization (WHO) for at least 1 year or confirmed negative C-peptide (<100pmol/l with concomitant blood glucose >4 mmol/l)
* Male subjects aged between 18-45 years
* HbA1c <8.0% (64mmol/mol) based on analysis from the central laboratory unit of the University Hospital Bern.
* Basal/Bolus-insulin regimen with insulin degludec for at least 3 months, with good knowledge of insulin self-management
* Regular physical activity (at least 30 min of moderate exercise 3 times weekly)
* Written informed consent

Exclusion Criteria:

* Relevant diabetic complications as judged by the investigator
* Total daily insulin dose >2 IU/kg/day
* Hypoglycaemia unawareness (Gold score > 4) or any episode of severe hypoglycaemia as defined by the American Diabetes Association within the last 6 months
* Physical or psychological disease likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator
* Current treatment with drugs known to interfere with metabolism, e.g. systemic corticosteroids, statins etc.
* Known fructose-intolerance or malabsorption
* Known allergy to one of the study drugs

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-08 (Actual)

PRIMARY OUTCOMES:
Time (in minutes) to hypoglycaemia (plasma glucose <3.9mmol/l) | From time point 0 minutes (initiation of exercise) to time point 60 minutes (completion of exercise) or development of hypoglycaemia
  The development of hypoglycaemia will be determined by repeated measurement of plasma glucose.

SECONDARY OUTCOMES:
Glucose levels before exercise | Time point -30 minutes until time point 0 minutes (initiation of exercise)
  Plasma glucose will be measured repeatedly every 5 minutes
Glucose levels during exercise | From time point 0 minutes until time point 60 minutes (completion of exercise) or development of hypoglycaemia
  Plasma glucose will be measured repeatedly every 5 minutes
Glucose levels after exercise | From time point 0 minutes until time point 90 minutes
  Plasma glucose will be measured repeatedly every 5 minutes
Lactate levels before exercise | From time point -30 minutes until time point 0 minutes (initiation of exercise)
  Lactate will be measured repeatedly every 5 minutes
Lactate levels during exercise | From time point 0 minutes until time point 60 minutes (completion of exercise) or development of hypoglycaemia
  Lactate will be measured repeatedly every 5 minutes
Lactate levels after exercise | From time point 0 minutes until time point 90 minutes
  Lactate will be measured repeatedly every 5 minutes
Insulin levels before exercise | Time point -30 minutes until time point 0 minutes (initiation of exercise)
  Lactate will be measured repeatedly every 15 minutes
Insulin levels during exercise | From time point 0 minutes until time point 60 minutes (completion of exercise) or development of hypoglycaemia
  Insulin will be measured repeatedly every 15 minutes
Insulin levels after exercise | From time point 0 minutes until time point 150 minutes
  Insulin will be measured repeatedly every 15 minutes
Heart rate before exercise | Time point -30 minutes until time point 0 minutes (initiation of exercise)
  Heart rate will be measured using an electro-cardio-gramme
Heart rate during exercise | From time point 0 minutes until time point 60 minutes (completion of exercise) or development of hypoglycaemia
  Heart rate will be measured using an electro-cardio-gramme
Oxygen consumption before exercise | Between 15 minutes and 5 minutes before initiation of exercise
  Oxygen consumption will be measured via spirometry
Oxygen consumption during exercise | Between 15 minutes and 20 minutes during exercise
  Oxygen consumption will be measured via spirometry
Carbon dioxide production before exercise | Between 15 minutes and 5 minutes before initiation of exercise
  Carbon dioxide production will be measured via spirometry
Carbon dioxide production during exercise | Between 15 minutes and 20 minutes during exercise
  Carbon dioxide production will be measured via spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Stettler, MD, Principal Investigator — Inselspital, Bern University Hospital, University of Bern
Locations (1):
- Division of Endocrinology, Diabetes and Clinical Nutrition, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kosinski C, Herzig D, Laesser CI, Nakas CT, Melmer A, Vogt A, Vogt B, Laimer M, Bally L, Stettler C. A Single Load of Fructose Attenuates the Risk of Exercise-Induced Hypoglycemia in Adults With Type 1 Diabetes on Ultra-Long-Acting Basal Insulin: A Randomized, Open-Label, Crossover Proof-of-Principle Study. Diabetes Care. 2020 Sep;43(9):2010-2016. doi: 10.2337/dc19-2250. Epub 2020 Jun 26. PMID 32591421